CLINICAL TRIAL: NCT03115723
Title: Frequency and Characteristics of Rehospitalizations During One Year After Percutaneous Coronary Intervention and Coronary Angiography - Results of the ACIRA Registry, Aquitaine Region
Brief Title: Analysis of Hospitalizations One Year After Acts of CAG and PCI in the Aquitaine région - ACIRA Register Data Analysis
Acronym: ACIRA-REHOSP
Status: Completed | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2014/29
Record Dates: First submitted 2017-04-10; First posted 2017-04-14 (Actual); Last update posted 2022-02-09 (Actual); Status verified 2022-02

CONDITIONS: Angioplasty; Coronary Angiography
Keywords: Hospitalization; Health Care Economics and Organizations
MeSH Terms: interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1 : Percutaneous coronary intervention: All the patients who underwent percutaneous coronary intervention, in 9 invasive cardiology centers in the Aquitaine Region, France.
  Interventions: Procedure: Percutaneous coronary intervention
- Group 2 : Coronary angiography: All the patients who underwent coronary angiography, in 9 invasive cardiology centers in the Aquitaine Region, France
  Interventions: Procedure: Coronary angiography

INTERVENTIONS:
Procedure: Percutaneous coronary intervention
  Groups: Group 1 : Percutaneous coronary intervention
Procedure: Coronary angiography
  Groups: Group 2 : Coronary angiography

SUMMARY:
Hospital readmission rate following percutaneous coronary interventions (PCI) or coronary angiographies (CAG) is a main indicator of quality of care and addresses economic issues. The aim of this study is to quantify the frequency and analyse the types of rehospitalizations and repeat revascularizations during one year after a PCI or a CAG. This information is needed to organize the health care pathway and to identify preventable rehospitalizations.

ELIGIBILITY:
Inclusion Criteria:

* Patients included in ACIRA Registry : All volunteer adults (≥ 18 years) and French resident patients who underwent PCI and CAG in the interventional cardiology hospitals in the Aquitaine region (France),
* Initial PCI or CAG performed from January 1, 2012 to December 31, 2013,
* Initial PCI or CAG performed in nine interventional cardiology hospitals in the Aquitaine region (France).

Exclusion Criteria:

* Patients who declined to take part of ACIRA Registry,
* Patients resident outside the Aquitaine region (France),
* Patients who died during the initial hospital stay,
* Patients hospitalized for a PCI or a CAG the month preceding the initial procedure including in the ACIRA-Rehosp study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All volunteer adults (≥ 18 years) and French resident patients who underwent PCI and CAG in nine interventional cardiology hospitals in the Aquitaine region (France), from January 1, 2012 to December 31, 2013.
Sampling Method: Non-Probability Sample
Enrollment: 11487 (Actual)
Dates: Start 2016-01-15 (Actual); Primary Completion 2017-01-15 (Actual); Study Completion 2017-01-15 (Actual)

PRIMARY OUTCOMES:
Type of rehospitalization | Baseline to 1 year
Number of rehospitalization | Baseline to 1 year

SECONDARY OUTCOMES:
Identification of hospitals | Baseline to 1 year
  All hospitals concerned by initial coverage and rehospitalization
Type of diagnoses and procedures associated with each type of rehospitalization | Baseline to 1 year
Type of cardiac rehabilitation procedures in hospitalizations for post-operative and rehabilitation wards | Baseline to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Saillour-Glénisson Florence, MD, Study Chair — University Hospital, Bordeaux; Lesaine Emilie, MD, Study Director — University Hospital, Bordeaux
Locations (11):
- France (11):
  - Clinique Esquirol St Hilaire, Agen
  - Clinique cardiologique d'Aressy, Aressy
  - GCS Bayonne, Bayonne
  - Clinique de Caudéran les pins-francs, Bordeaux
  - Clinique de St Augustin, Bordeaux
  - CH de Libourne, Libourne
  - CH de Mont de Marsan, Mont-de-Marsan
  - CH de Pau, Pau
  - CHU de Bordeaux, Pessac
  - Hôpital privé St Martin, Pessac
  - CH de Perigueux, Périgueux

IPD SHARING:
Plan to Share IPD: No